CLINICAL TRIAL: NCT00676442
Title: An Open-Label, Randomized, Four-Way Crossover Study to Evaluate the Effect of Food on the Bioavailability of Naproxen and Esomeprazole From a PN 400 Tablet in Healthy Subjects
Brief Title: Study Evaluating the Effect of Food on the Bioavailability of PN400 Components
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: POZEN (Industry)
Responsible Party: Director, Clinical Research, Pozen
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: PN400-103
Record Dates: First submitted 2008-05-08; First posted 2008-05-13 (Estimated); Last update posted 2008-09-05 (Estimated); Status verified 2008-09

CONDITIONS: Arthritis
MeSH Terms: conditions — Arthritis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- 1 (Other): PN400 administered after meal
  Interventions: Drug: PN400
- 2 (Other): PN400 administered prior to meal
  Interventions: Drug: PN400
- 3 (Other): PN400 administered prior to meal
  Interventions: Drug: PN400
- 4 (Other): PN400 followed by fast
  Interventions: Drug: PN400

INTERVENTIONS:
Drug: PN400 — naproxen/esomeprazole

SUMMARY:
We will evaluate the effect of food on the bioavailability of the components of PN400

ELIGIBILITY:
Inclusion Criteria:

* Healthy male or non-pregnant female subjects between 18-55 years old as well as other standard inclusion criteria for a study of this nature.

Exclusion Criteria:

* Standard exclusion criteria for a study of this nature.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2008-05; Primary Completion 2008-06 (Actual); Study Completion 2008-06 (Actual)

PRIMARY OUTCOMES:
To determine the effects of food eaten at different times on the bioavailability of the components of PN400 following a single oral dose in healthy subjects. | 72-hours

SECONDARY OUTCOMES:
To assess the safety and tolerability of PN 400 under fasting and fed conditions. | entire study duration

CONTACTS AND LOCATIONS:
Locations (1):
- Austin, Texas, United States